CLINICAL TRIAL: NCT01356030
Title: Prospective Comparison of EUS-guided FNA and ERCP Tissue Sampling for the Diagnosis of Suspected Pancreato-biliary Neoplasms
Brief Title: Endoscopic Ultrasound Versus Endoscopic Retrograde Cholangiopancreatography (ERCP) Tissue Sampling for the Diagnosis of Suspected Pancreatico-Biliary Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Pacific Medical Center Research Institute (Other)
Responsible Party: Principal Investigator, Janak Shah, MD, Director of Pancreatic and Biliary Endoscopy, California Pacific Medical Center Research Institute
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2011.048
Record Dates: First submitted 2011-05-12; First posted 2011-05-19 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Pancreaticobiliary Cancers; Jaundice; Bile Duct Obstruction
MeSH Terms: conditions — Jaundice; Cholestasis | interventions — Cholangiopancreatography, Endoscopic Retrograde; Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- EUS-FNA (Active Comparator)
  Interventions: Procedure: EUS FNA
- ERCP Brushing and Biopsy (Active Comparator)
  Interventions: Procedure: ERCP

INTERVENTIONS:
Procedure: ERCP — Endoscopic retrograde cholangiopancreatography (ERCP) is usually clinically indicated to place a stent (a plastic or metal tube) in the bile duct. The ERCP procedure is an endoscopic exam during which a small catheter or wire is placed into the bile duct from the point at which it connects to the small intestine. During such a procedure a stent can then be placed to help drain the bile across the site of blockage, and thereby treat your jaundice.
  Arms: ERCP Brushing and Biopsy
Procedure: EUS FNA — Endoscopic ultrasound (EUS) is a procedure in which a flexible tube with a tiny camera and ultrasound probe at the tip is placed through the mouth, down the esophagus, and into the stomach and duodenum (first part of the small intestine where bile flows from the bile duct into the intestine). This allows the doctor performing the EUS to get a much closer view of your pancreas and bile duct. If a suspicious mass is seen, a small sample of the mass (biopsy) is taken using fine needle aspiration (FNA). FNA involves the use of a thin hollow needle to extract cells for diagnostic purposes and is considered safer and less invasive than surgical biopsies.
  Arms: EUS-FNA

SUMMARY:
The two most commonly used methods to biopsy suspected pancreaticobiliary masses are (1) endoscopic ultrasound guided fine-needle aspiration (EUS-FNA) and (2) cytology brush biopsies obtained during endoscopic retrograde cholangiopancreatography (ERCP). At most centers, the specific method used depends on the availability of the technology and local expertise. Although it is believed that EUS-FNA is more accurate than ERCP brushings, there have been no head-to-head comparisons. The investigators' hypothesis is that EUS-FNA is superior to ERCP in obtaining tissue biopsies of pancreaticobiliary tumors, and the investigators aim to directly compare the two techniques.

DETAILED DESCRIPTION:
Patients with pancreaticobiliary tumors usually present with painless jaundice due to bile duct obstruction. The standard clinical evaluation may include EUS and/or ERCP. At centers where EUS is available (like CPMC), it is usually used first as it is generally considered a better tool for tumor detection, staging, and performing biopsies (FNA). ERCP is then performed, if needed, to place a stent and relieve jaundice. As EUS is a relatively newer technology that has not widely disseminated, other centers use ERCP as the 1st modality to evaluate suspected malignant pancreaticobiliary obstruction. The role of ERCP in this setting is to not only place a stent to relieve jaundice, but to additionally obtain cytology brushings for tissue diagnosis.

Several studies have reported high sensitivity of EUS-FNA for detecting pancreaticobiliary cancers that are causing bile duct obstruction and jaundice (80-90%). The sensitivity for ERCP brushings and biopsies to detect the same types of tumors is reportedly lower (30-80%), but there have been no direct comparisons of these techniques.

Few centers use both technologies (EUS and ERCP) for patient care, or often perform EUS and ERCP at separate sessions. At CPMC, the investigators routinely perform EUS and ERCP together for patients needing these procedures. Thus the investigators are in a unique position to directly compare EUS-FNA to ERCP brushings for tissue diagnosis of suspected pancreaticobiliary tumors.

The proposed study will be the 1st direct comparison of EUS-FNA to ERCP tissue sampling for patients with suspected pancreaticobiliary cancers. Study results will highlight the best approach to obtain a biopsy diagnosis of pancreatic and biliary tract cancers.

ELIGIBILITY:
Inclusion Criteria:

* Patients age >18 years that are scheduled for EUS and possible ERCP for the evaluation of jaundice from suspected pancreaticobiliary tumors.

Exclusion Criteria:

* Patients that do not provide consent for EUS and ERCP (for standard clinical reasons)
* Patients that do not require ERCP based on EUS findings (e.g. no mass seen, mass is not causing jaundice
* Patients in whom an additional 5 minutes of procedure time may increase the procedural/sedation risks:

  * pregnant patients
  * patients with severe medical co-morbidities (ASA class 4 or 5)
* Patients with significant bleeding risk precluding endoscopic tissue sampling

  * INR > 1.4 or Prothrombin time > 5 sec more than control
  * Platelet count < 50,000

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Direct comparison of tissue sampling techniques for patients with suspected pancreaticobiliary cancers. | One year
  Diagnostic yield from EUS-FNA samples will be compared to yield from ERCP tissue sampling methods (brushings and forceps biopsies).

CONTACTS AND LOCATIONS:
Overall Officials: Janak Shah, MD, Principal Investigator — California Pacific Medical Center
Locations (1):
- California Pacific Medical Center, San Francisco, California, United States

REFERENCES:
- [Background] Larghi A, Waxman I. Differentiating benign from malignant idiopathic biliary strictures: are we there yet? Gastrointest Endosc. 2007 Jul;66(1):97-9. doi: 10.1016/j.gie.2006.12.047. No abstract available. PMID 17591480
- [Background] Hollerbach S. EUS and ERCP: brothers in arms. Gastrointest Endosc. 2008 Sep;68(3):467-9. doi: 10.1016/j.gie.2008.01.022. No abstract available. PMID 18760174
- [Background] Ross WA, Wasan SM, Evans DB, Wolff RA, Trapani LV, Staerkel GA, Prindiville T, Lee JH. Combined EUS with FNA and ERCP for the evaluation of patients with obstructive jaundice from presumed pancreatic malignancy. Gastrointest Endosc. 2008 Sep;68(3):461-6. doi: 10.1016/j.gie.2007.11.033. Epub 2008 Apr 2. PMID 18384788
- [Background] Savides TJ, Donohue M, Hunt G, Al-Haddad M, Aslanian H, Ben-Menachem T, Chen VK, Coyle W, Deutsch J, DeWitt J, Dhawan M, Eckardt A, Eloubeidi M, Esker A, Gordon SR, Gress F, Ikenberry S, Joyce AM, Klapman J, Lo S, Maluf-Filho F, Nickl N, Singh V, Wills J, Behling C. EUS-guided FNA diagnostic yield of malignancy in solid pancreatic masses: a benchmark for quality performance measurement. Gastrointest Endosc. 2007 Aug;66(2):277-82. doi: 10.1016/j.gie.2007.01.017. PMID 17643700
- [Background] Sanchez MV, Pujol B, Napoleon B. Linear array EUS in bile-duct lesions. Gastrointest Endosc. 2009 Feb;69(2 Suppl):S121-4. doi: 10.1016/j.gie.2008.12.016. No abstract available. PMID 19179135
- [Background] Fogel EL, deBellis M, McHenry L, Watkins JL, Chappo J, Cramer H, Schmidt S, Lazzell-Pannell L, Sherman S, Lehman GA. Effectiveness of a new long cytology brush in the evaluation of malignant biliary obstruction: a prospective study. Gastrointest Endosc. 2006 Jan;63(1):71-7. doi: 10.1016/j.gie.2005.08.039. PMID 16377319
- [Background] de Bellis M, Sherman S, Fogel EL, Cramer H, Chappo J, McHenry L Jr, Watkins JL, Lehman GA. Tissue sampling at ERCP in suspected malignant biliary strictures (Part 2). Gastrointest Endosc. 2002 Nov;56(5):720-30. doi: 10.1067/mge.2002.129219. No abstract available. PMID 12397282
- [Background] Fritscher-Ravens A, Broering DC, Knoefel WT, Rogiers X, Swain P, Thonke F, Bobrowski C, Topalidis T, Soehendra N. EUS-guided fine-needle aspiration of suspected hilar cholangiocarcinoma in potentially operable patients with negative brush cytology. Am J Gastroenterol. 2004 Jan;99(1):45-51. doi: 10.1046/j.1572-0241.2003.04006.x. PMID 14687140
- [Background] Eloubeidi MA, Chen VK, Jhala NC, Eltoum IE, Jhala D, Chhieng DC, Syed SA, Vickers SM, Mel Wilcox C. Endoscopic ultrasound-guided fine needle aspiration biopsy of suspected cholangiocarcinoma. Clin Gastroenterol Hepatol. 2004 Mar;2(3):209-13. doi: 10.1016/s1542-3565(04)00005-9. PMID 15017604
- [Background] DeWitt J, Misra VL, Leblanc JK, McHenry L, Sherman S. EUS-guided FNA of proximal biliary strictures after negative ERCP brush cytology results. Gastrointest Endosc. 2006 Sep;64(3):325-33. doi: 10.1016/j.gie.2005.11.064. PMID 16923477
- [Background] Rosch T, Hofrichter K, Frimberger E, Meining A, Born P, Weigert N, Allescher HD, Classen M, Barbur M, Schenck U, Werner M. ERCP or EUS for tissue diagnosis of biliary strictures? A prospective comparative study. Gastrointest Endosc. 2004 Sep;60(3):390-6. doi: 10.1016/s0016-5107(04)01732-8. PMID 15332029
- [Background] Lee JH, Salem R, Aslanian H, Chacho M, Topazian M. Endoscopic ultrasound and fine-needle aspiration of unexplained bile duct strictures. Am J Gastroenterol. 2004 Jun;99(6):1069-73. doi: 10.1111/j.1572-0241.2004.30223.x. PMID 15180727
- [Background] Uehara H, Tatsumi K, Masuda E, Kato M, Kizu T, Ishida T, Takakura R, Takano Y, Nakaizumi A, Ishikawa O, Takenaka A. Scraping cytology with a guidewire for pancreatic-ductal strictures. Gastrointest Endosc. 2009 Jul;70(1):52-9. doi: 10.1016/j.gie.2008.09.059. Epub 2009 Feb 26. PMID 19249043
- [Background] DeWitt J, McGreevy K, Sherman S, LeBlanc J. Utility of a repeated EUS at a tertiary-referral center. Gastrointest Endosc. 2008 Apr;67(4):610-9. doi: 10.1016/j.gie.2007.09.037. Epub 2008 Feb 14. PMID 18279866
- [Derived] Weilert F, Bhat YM, Binmoeller KF, Kane S, Jaffee IM, Shaw RE, Cameron R, Hashimoto Y, Shah JN. EUS-FNA is superior to ERCP-based tissue sampling in suspected malignant biliary obstruction: results of a prospective, single-blind, comparative study. Gastrointest Endosc. 2014 Jul;80(1):97-104. doi: 10.1016/j.gie.2013.12.031. Epub 2014 Feb 19. PMID 24559784